CLINICAL TRIAL: NCT06262932
Title: Effectiveness of Repeated Amiodarone Dosing Regimen Versus Standard Dosing Regimen in Atrial Fibrillation Patient With Rapid Ventricular Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Police General Hospital, Thailand (Other)
Responsible Party: Principal Investigator, Chawit Lopimpisuth, Principal Investigator, Police General Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADS regimen
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeated amiodarone bolus dosing regimen (Active Comparator): An Initial 150 mg IV amiodarone bolus should be given over a 15-minute period. If the heart rate is still over 110 minutes after the initial treatment, provide an additional 150 mg IV amiodarone bolus over a 15-minute period. During the first 24 hours, this bolus may be administered up to three times in total. Within 24 hours of finishing the first bolus dosage, 900 mg of amiodarone will be administered intravenously.
  Interventions: Drug: Amiodarone
- Standard dosing regimen (Active Comparator): An Initial 150 mg IV amiodarone bolus should be given over a 15-minute period, then a 24-hour amiodarone loading infusion 900 mg over 24 hours
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Amiodarone — Assess the effectiveness of repeated bolus dosing strategies of amiodarone.

SUMMARY:
The goal of this clinical trial is to compare in atrial fibrillation patient with rapid ventricular response. The main question it aims to answer are Effectiveness of Repeated Amiodarone dosing regimen versus standard dosing regimen in Atrial fibrillation patient with rapid ventricular response Participants will receive Amiodarone iv treatment with different regimen

* Repeated dosing regimen
* Standard dosing regimen

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* Atrial fibrillation with rapid ventricular response patient (ventricular rate > 110)

Exclusion Criteria:

* Baseline EKG Corrected QT interval (QTc) < 500 msec
* History of pulmonary fibrosis
* History of Cirrhosis
* Cardiac Index <2.2 L/min/m2 or Cardiogenic shock
* Unstable arrhythmia
* Receive amiodarone within 3 months prior to present illness
* Pregnancy
* Amiodarone or Iodine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Heart rate | 6-hours after receiving amiodarone bolus
  Percentage of patients who have Atrial fibrillation with rapid ventricular response, the percentage of patients who have heart rate below 110 bpms at 6 hours after receiving a repeated amiodarone bolus and loading dose regimen to the percentage of patients who have heart rate below 110 bpms at 6 hour after a conventional amiodarone IV loading dose regimen

SECONDARY OUTCOMES:
Normal sinus rhythm at 24 hours | 24-hours after receiving amiodarone bolus
  Percentage of patients who develop Atrial fibrillation with rapid ventricular response, the percentage of patients who have converted to sinus rhythm at 24-hours after receiving a repeated amiodarone bolus and loading dose regimen to the percentage of patients who have converted to sinus rhythm after a conventional amiodarone IV loading dose regimen
Heart rate | 24-hours after receiving amiodarone bolus
  Percentage of patients who have Atrial fibrillation with rapid ventricular response, the percentage of patients who have heart rate below 110 bpms at 24 hours after receiving a repeated amiodarone bolus and loading dose regimen to the percentage of patients who have heart rate below 110 bpms at 6 hour after a conventional amiodarone IV loading dose regimen
Major adverse cardiovascular events | 30 days after receiving amiodarone bolus
  Number of MACE [MACE defined as acute myocardial infarction (AMI), stroke, or cardiovascular death]
Phlebitis | 24-hours after receiving amiodarone bolus
  Rate of phlebitis complication during amiodarone infusion
Changed in heart rate | 24-hours after receiving amiodarone bolus
  Compare number of total heart rate induction in patients who received a repeated amiodarone bolus and loading dose regimen and a conventional amiodarone IV loading dose regimen at 24 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Police general hospital, Bangkok, Thailand